CLINICAL TRIAL: NCT01034826
Title: Progression to Impaired Glucose Tolerance and Type 2 Diabetes in the Korean People-based KNDP Study
Status: Completed | Type: Observational
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Korea university Guro Hospital Endocrinology department, Korea university
Other Study IDs: KNDP IGT study
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2009-12

CONDITIONS: Impaired Glucose Tolerance; Diabetes
Keywords: NGT, IGT, diabetes
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- life style modification: everyone in this study was advised about their life style, diet, exercise habits.

SUMMARY:
Impaired glucose tolerance is a metabolic state between normal glucose homeostasis and diabetes. Previously, prospective studies have shown higher progression rates from IGT to diabetes in other country. But There is no prospective-multicenter based reports in Korea. Therefore, the purpose of this study is to estimate the progression rates to impair glucose regulation and diabetes in the Korean population-based Korea national Diabetes program.

ELIGIBILITY:
Inclusion Criteria:

* fastic serum glucose >100 and/or pp2 serum glucose <200

Exclusion Criteria:

* known diabetes
* organ failure(For example, liver, kidney)
* known malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who vist the endocrinology department due to impaired fasting glucose or impaired glucose tolerance, or both.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
fasting serum glucose, fasting plasma insulin,post prandial serum glucose, post prandial plasma insulin, hbA1c | 0.1.3.5 year

REFERENCES:
- [Derived] Choi KM, Hwang SY, Hong HC, Yang SJ, Choi HY, Yoo HJ, Lee KW, Nam MS, Park YS, Woo JT, Kim YS, Choi DS, Youn BS, Baik SH. C1q/TNF-related protein-3 (CTRP-3) and pigment epithelium-derived factor (PEDF) concentrations in patients with type 2 diabetes and metabolic syndrome. Diabetes. 2012 Nov;61(11):2932-6. doi: 10.2337/db12-0217. Epub 2012 Jul 26. PMID 22837306